CLINICAL TRIAL: NCT02759211
Title: Pilot Trial of Backwards Walking in Persons With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Rehabilitation Hospital (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Jennifer Ruiz, DPT, Research Manager, Mandell Center for Multiple Sclerosis, Mount Sinai Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFH-16-27
Record Dates: First submitted 2016-03-22; First posted 2016-05-03 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Forwards Walking Group (FWG) (Active Comparator): The intervention will consist of three (3), treadmill exercise sessions per week, for eight (8) weeks, for a total of 24 exercise sessions.
  Interventions: Other: Forwards Walking
- Backwards Walking Group (BWG) (Experimental): The intervention will consist of three (3), treadmill exercise sessions per week, for eight (8) weeks, for a total of 24 exercise sessions.
  Interventions: Other: Backwards Walking

INTERVENTIONS:
Other: Backwards Walking — The Backwards Walking Group will perform backwards walking for the entire treatment intervention.
  Arms: Backwards Walking Group (BWG)
Other: Forwards Walking — The Forwards Walking Group will perform forwards walking for the entire treatment intervention.
  Arms: Forwards Walking Group (FWG)

SUMMARY:
There have been no published studies to date on the effects of backwards walking in persons with MS. Thus it is important that the investigators explore different methods for treatment to help improve balance and gait and prevent injury in persons with MS with gait disturbances and balance impairments.The overall goal of this research is to collect pilot data on the effectiveness of backwards walking as a therapy for improving spatiotemporal, clinical gait and balance assessments in persons with Multiple Sclerosis compared to forward walking.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of MS
* Cognitively able to understand directions and complete protocol (score of 22 or greater on MMSE)
* Signed Consent form approved by the Saint Francis Institutional Review Board
* 18-65 years of age
* PDDS score of 3 to 5 during the past 12 months
* Completion of the 6 minute walk test
* Speaks English (in order to safely complete intervention)

Exclusion Criteria:

* Unwilling or unable to complete assessments and intervention
* Current participation in physical therapy
* Major changes in exercise habits in the past three months
* Has had a relapse, acute Solumedrol treatment, or Acthar treatment in the past two months
* Requires constant bilateral assistance (canes or crutches) for ambulation and/or cannot walk at least 100 meters without resting
* Current self-reported medical history of unstable angina, uncontrolled cardiac dysrhythmias causing symptoms, symptomatic severe aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus or pulmonary infarction, history of DVT, acute myocarditis or pericarditis, acute systemic infection, uncontrolled hypertension, and uncontrolled diabetes [11]
* Participants that cannot adhere to the protocol, have an abnormal response to exercise, or is determined to be unsafe may be withdrawn at the discretion of the Principal Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Spatiotemporal Walking Parameters from Gaitrite Mat | Change in Baseline Spatiotemporal Walking parameters from Gaitrite Mat after 8 week intervention
  Change in Baseline Spatiotemporal Walking parameters from Gaitrite Mat after 8 week intervention
Gait Speed (Timed 25 Foot Walk) | Change in f Baseline Gait Speed (Timed 25 Foot Walk) after 8 week intervention
  Timed 25 Foot Walk
Single Leg Stance (SLS) | Change in Baseline SLS after 8 week intervention

SECONDARY OUTCOMES:
Timed-up and Go | Change in Baseline TUG after 8 week intervention
Activities-Specific Balance Confidence Scale (ABC) | Change in Baseline ABC after 8 week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Mandell Center for Multiple Sclerosis at the Mount Sinai Rehabilitation Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No